CLINICAL TRIAL: NCT01463241
Title: Behavioral and Affective Skills in Coping: Practice-Adapted Child Psychotherapy
Brief Title: Behavioral and Affective Skills in Coping (BASIC) Open Trial
Acronym: BASIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Judge Baker Children's Center (Other)
Responsible Party: Principal Investigator, John R. Weisz, PhD, ABPP, Professor of Psychology, Harvard University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R34MH085963-03 (NIH)
Record Dates: First submitted 2011-10-26; First posted 2011-11-01 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Anxiety Disorders; Depressive Disorders; Disruptive Behavior Disorders
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Attention Deficit and Disruptive Behavior Disorders | interventions — Coping Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BASIC treatment (Other): As an open trial, all participants in this study will receive the BASIC treatment.
  Interventions: Behavioral: Behavioral and Affective Skills in Coping (BASIC)

INTERVENTIONS:
Behavioral: Behavioral and Affective Skills in Coping (BASIC) — The investigator's seek to develop a treatment protocol that integrates five core intervention principles that are common to evidence-based treatments for youth depression, anxiety, and disruptive behavior problems. The protocol will be designed for implementation in everyday community practice settings by practitioners. The BASIC protocol will include (a) a therapist manual guiding the use of five BASIC skills [Belief Repair, Action, Solving Problems, Incentives, and Calming]; (b) child and parent materials to facilitate learning skills, practicing them in-session, and using them outside sessions; and (c) a decision tree to guide judgments about which skills to use and when to switch skills or treatment focus.

SUMMARY:
The overall objective of the project is to develop and assess the feasibility of a brief, practice-friendly approach to psychotherapy for children, entitled Behavioral and Affective Skills in Coping (BASIC) and designed for use as a first step toward evidence-based practice by practitioners in clinical service settings.

DETAILED DESCRIPTION:
The investigators seek to develop a treatment protocol that integrates five core intervention principles that are common to evidence-based treatments for youth depression, anxiety, and disruptive behavior problems. The protocol will be designed for implementation in everyday community practice settings by practitioners. Because many empirically supported treatments for youth disorders address only one area of impairment, they may not be an ideal fit to community clinics, where (a) most practitioners treat an array of disorders rather than specializing in just one, (b) most referred youths present with multiple disorders, and (c) priority problems and treatment needs may shift for many youths during an episode of care. Moreover, because many evidence-based treatments have been developed in research settings, they may not be designed in ways that are ideal for front-line therapists in community settings. The investigators hope to reduce the difficulty of transporting treatments into community practice by incorporating the perspectives of community practitioners in the development and design of the protocol. By incorporating the feedback of expert treatment developers, the investigators hope to ensure that BASIC is not only appealing to users but also consistent with what has been learned through treatment research over the years. Finally, the trial will provide preliminary evidence on whether this brief "first course" in evidence-based treatment is beneficial for youths with depression, anxiety, and disruptive behavior problems-three clusters that account for a large percentage of youth referrals.

ELIGIBILITY:
Inclusion Criteria:

* 8-15 year-old youth
* The youth will meet diagnostic criteria for one or more target disorders in the broad areas of anxiety (including Generalized Anxiety Disorder, Separation Anxiety Disorder, Social Phobia, Obsessive Compulsive Disorder, Specific Phobia, Panic Disorder, Anxiety Disorder Not Otherwise Specified, Adjustment Disorder with Anxiety), depression (including Major Depressive Disorder, Dysthymic Disorder, Minor Depression, Depressive Disorder Not Otherwise Specified, Adjustment Disorder with Depressed Mood), and conduct (Oppositional Defiant Disorder, Conduct Disorder, Disruptive Behavior Disorder Not Otherwise Specified, Adjustment Disorder with Disturbance of Conduct).

Exclusion Criteria:

* Youth with primary ADHD
* Youth with developmental disorders
* Youth with symptoms of a thought disorder including delusions and hallucinations

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2011-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in diagnostic status at post-treatment: Schedule for Affective Disorders and Schizophrenia for School-Age Children- Present and Lifetime Version (K-SADS-PL) | Immediately before and after the treatment course, which is expected to last an average of 7 months
  The K-SADS-PL (Puig-Antich & Chambers, 1983; Kaufman et al., 1997) is a semi-structured diagnostic interview designed to be used for youth ages 6 through 18. The K-SADS-PL will be used to diagnose DSM-IV disorders, and has been found to have acceptable test-retest reliability (κs = .60 - 1.00), inter-rater reliability (κs = .60 - 1.00) and internal consistency (αs = .68 - .84), and to discriminate between disordered and non-disordered children (Ambrosini, 2000; Kaufman et al., 1997; Lewinsohn, et al., 1994).
Change from baseline in child/adolescent problem areas at post-treatment: Child Behavior Checklist -- Problem Portion (CBCL) | Immediately before and after the treatment course, which is expected to last an average of 7 months
  The CBCL obtains caregiver reports on 118 child/adolescent problems, each rated on a 0-1-2 scale. The CBCL is a widely-used and psychometrically sound measure with well-developed norms (Achenbach, 2001), and it yields T-scores for eight narrow-band syndrome scales (Anxious-Depressed, Withdrawn-Depressed, Somatic Complaints, Attention Problems, Thought Problems, Social Problems, Aggressive Behavior, and Rule-Breaking Behavior), two broad-band second-order syndrome scales (Internalizing and Externalizing), and a Total Problems scale.
Change from baseline in child/adolescent problem areas at post-treatment: Youth Self-Report Form -- Problem Portion (YSR) | Immediately before and after the treatment course, which is expected to last an average of 7 months
  The YSR is a 118-items assessing symptoms across a broad range of clinical significance, overlapping heavily with the content of the parent-report CBCL. The YSR is normed for children aged 11 and older, but item wording is quite simple, and data from clinic-referred children (Yeh & Weisz, 2001) have shown that the measure performs as well psychometrically for children aged 7-10 as for youths aged 11-17; this suggests that the YSR may be appropriately employed with youngsters across the full age range of the current sample.
Change from baseline in child/adolescent problem areas during treatment and at post-treatment: Brief Problem Checklist (BPC; Chorpita, Reise, Weisz, et al. 2010) | Participants will be followed for the duration of the treatment course, an expected average of 7 months
  The BPC is a 12-item questionnaire that has both parent and youth versions designed to provide a brief, easily administered, clinically relevant, and psychometrically sound measure of symptoms and problems. The items for this measure were developed using item response theory and factor analysis applied to the CBCL and YSR and ask about symptoms of internalizing and externalizing problems in the last week. Internal consistency for the BPC ranged from .70 to .83. Test-retest reliability was also good, with Cronbach's alpha falling in the range of .72 to.79.
Change from baseline in target problem during treatment and at post-treatment: Weekly Target Problem Report (TPR; STEPs Team, 2008) | Participants will be followed for the duration of the treatment course, an expected average of 7 months
  The TPR tracks trajectories of change in the target problems identified by caregivers and children at the start of treatment. In the initial assessment, the caregiver and child are separately asked to identify the "problems for which you/your child most need/s help." The 3 top-ranked problems are then rated for severity in weekly phone calls. TPR ratings have been shown to be sensitive to change over time and in ways that differ for different treatments; moreover, the TPR is a consumer-sensitive index of treatment response, reflecting the concerns for which caregiver and child sought help.
Change from baseline in clinical global impression during treatment course: Clinical Global Impression-Improvement (CGI-I) Scale (Guy, 1970). | Participants will be followed for the duration of the treatment course, an expected average of 7 months
  The CGI-I is a 7-point scale to be completed by practitioners each week, indicating their rating of client improvement relative to baseline severity. The CGI-I has been used as a measure of treatment response in studies testing CBT for anxiety disorders, CBT for depression, and Behavioral Caregiver Training for disruptive behavior in children with ADHD. The CGI-I has demonstrated acceptable convergent validity between clinicians and blind assessors rating children's response to treatment.

SECONDARY OUTCOMES:
Services for Children & Adolescents - Parent Interview (SCAPI; Jensen et al., 2004) | Participants will be followed for the duration of the treatment course, an expected average of 7 months
  The SCAPI is an interview administered to parents to assess children's services use across primary care, specialty mental health, and other settings. It is administered in two parts. In Part I, parents are asked about psychotropic medications the child receives. In Part II, parents are asked to document any recent visits the child has made to their physician. Test-retest κ values ranged from .49 to 1.00, with an overall κ value for all services of .97.
Service Assessment for Children and Adolescents-Treatment and Auxiliary Service Use Scales (SACA; Horwitz et al., 2001) | Participants will be followed for the duration of the treatment course, an expected average of 7 months
  The SACA is a standardized interview for parents that collects information on use of mental health services across a broad spectrum (including outpatient, inpatient, and school-based). SACA reliability and validity data are well-documented.
Therapeutic Alliance Scale for Children (TASC; Shirk & Saiz, 1992) | Following the participant's treatment course, which is expected to last an average of 7 months
  The TASC assesses the quality of youths' working alliance with their therapists. Originally designed to examine youth in inpatient settings, the 9-item revised scale comes in both a youth-report form and a parent-report form (parents reporting on their youth's relationship with the therapist). The TASC has demonstrated adequate internal consistency ranging from .72 to .74.
Therapy Process Observational Coding System-Alliance Scale (TPOCS-A; McLeod & Weisz, 2005) | Following the participant's treatment course, which is expected to last an average of 7 months
  The TPOCS-A assesses child-clinician and caregiver-clinician alliance through observational ratings of recorded therapy sessions. The TPOCS-A was derived from questionnaire measures of alliance, adapting items that could be expressed in terms of observable behavior, both reflecting alliance or its absence. Psychometric analyses based on child and caregiver sessions in community outpatient clinics showed that both child and caregiver forms have good inter-rater reliability and internal consistency. Psychometric analyses also found that both child and caregiver forms predicted treatment outcome.
Parent Child Satisfaction Scales (PCSS; Hawley, Weersing, & Weisz, 1998) | Following the participant's treatment course, which is expected to last an average of 7 months
  The Parent Child Satisfaction Scales consist of an 8-item parent measure and an 8-item child measure that assess the child's satisfaction with the treatment he or she received as well as the parents' satisfaction with their child's treatment.
Therapist Satisfaction Inventory (TSI; Addis & Krasnow's, 2000) | Following the clinician's participation in the study, which is anticipated to last 18 months
  The TSI is a 16-item therapist-report measure derived from Addis & Krasnow's (2000) report on therapist attitudes toward manualized treatments. The items encompass whether therapists liked the treatment approach they used, whether they perceived that the approach was effective, whether they believe it allowed them to individualize treatment to fit client needs, and whether the approach seems appropriate for the kinds of children they most often see.

CONTACTS AND LOCATIONS:
Overall Officials: John R Weisz, Ph.D., ABPP, Principal Investigator — Department of Psychology, Harvard University
Locations (1):
- Judge Baker Children's Center, Boston, Massachusetts, United States